CLINICAL TRIAL: NCT03610178
Title: Genetic and Epigenetic Mechanisms of Developing Gestational Diabetes Mellitus and Its Effects on the Fetus: a Randomised Controlled Trial of Different Glycemic Targets During Pregnancy
Brief Title: Genetic and Epigenetic Mechanisms of Developing Gestational Diabetes Mellitus and Its Effects on the Fetus
Acronym: GEM GDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-14-30012
Record Dates: First submitted 2017-11-13; First posted 2018-08-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Women with GDM are randomised to 2 treatment groups: group 1 - treatment group with very tight glycemic targets (<5.1 mmol / L fasting glucose and <7.0 mmol / l hour after a meal) and group 2 - treatment group with tight-moderate glycemic targets (<5.3 mmol / L fasting glucose and <7.8 mmol / l in an hour after a meal).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- very tight glycemic targets (Active Comparator)
  Interventions: Other: Very tight glycemic targets, life-style modification, insulin therapy if needed
- tight-moderate glycemic targets (Active Comparator): Less tight glycemic targets
  Interventions: Other: Tight-moderate glycemic targets, life-style modification, insulin therapy if needed
- Control group (No Intervention): Only observation in women with normal glucose tolerance

INTERVENTIONS:
Other: Very tight glycemic targets, life-style modification, insulin therapy if needed — All patients are assigned to life-style modification (diet and physical exercise). If target glucose levels (<5.1 mmol/L fasting and <7.0 mmol/L postprandial) are not achieved insulin therapy is started
  Other Names: Tight glycemic targets
  Arms: very tight glycemic targets
Other: Tight-moderate glycemic targets, life-style modification, insulin therapy if needed — All patients are assigned to life-style modification (diet and physical exercise). If target glucose levels (<5.3 mmol/L fasting and <7.8 mmol/L postprandial) are not achieved insulin therapy is started
  Arms: tight-moderate glycemic targets

SUMMARY:
This is a randomized controlled trial of different glycemic targets during tratment of women with GDM with assessement of epygenetic aspects of their effects on the fetus and pregnancy outcomes. This study is interventional, randomised controlled trial, open-label.

DETAILED DESCRIPTION:
The study aims to clarify the effect of hyperglycemia and its correction, the level of physical activity and consumption of major macro- and micronutrients by women during pregnancy on DNA methylation and expression of genes involved in neuroendocrine regulation and development of metabolic diseases in offspring, as well as functional characteristics of human umbilical vein endothelial cells (HUVECs). For the purpose of the study women with GDM are randomised to 2 treatment groups per glycemic targets ( very tight and tight-moderate glycemic targets). Data on glycenmic levels during the study and consumption of major macro- and micronutrients will be collected using a mobile application with electronic dairies report forms.

This clinical trial record primarily describes the overarching observational cohort study "Genetic and Epigenetic Mechanisms of Developing Gestational Diabetes Mellitus and Its Effects on the Fetus" including women with GDM and healthy pregnant women.

Substudy Protocol: A key predefined component of this larger study is an interventional, randomized controlled substudy entitled "Tight versus less tight glycaemic targets for women with gestational diabetes mellitus: a randomised controlled trial" (also known as the GEM GDM Trial).

The GEM GDM Trial is an open-label, randomized controlled trial (RCT) that compares the effects of tight (very tight) versus less tight (tight-moderate) glycemic control on maternal and neonatal outcomes in women diagnosed with Gestational Diabetes Mellitus (GDM). Participants from the main GEM cohort who are diagnosed with GDM according to International Association of the Diabetes and Pregnancy Study Groups (IADPSG) criteria are eligible for screening and subsequent randomization into this substudy.

The substudy aims to enroll 650 pregnant women with a singleton pregnancy and GDM, randomly assigning them in a 1:1 ratio to one of two glycemic target groups.

* Tight Target Group: Fasting capillary glucose <5.1 mmol/L (<92 mg/dL); 1-hour postprandial glucose <7.0 mmol/L (<126 mg/dL).
* Less Tight Target Group: Fasting capillary glucose <5.3 mmol/L (<95 mg/dL); 1-hour postprandial glucose <7.8 mmol/L (<140 mg/dL).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with GDM diagnosed according to the Russian national consensus and the recommendations of the International Association of Diabetes and Pregnancy Study Groups (fasting glucose of ≥5.1 mmol/L, and/or ≥10.0 mmol/L after 1 h, and/or ≥8.5 mmol/L after 2 h in oral glucose tolerance test (OGTT) with 75 g of glucose).
* Gestational age at the time of inclusion in the study 12 weeks 0 days - 31 weeks 6 days
* For control group: pregnant women with normal glucose tolerance confirmed by OGTT at 24-31 weeks of gestation.

Exclusion Criteria:

* Diabetes mellitus type 1 and tipe 2
* Other deseases that affect methabolism of carbohydrates
* Use of drugs that affect methabolism of carbohydrates
* Malformations of the fetus identifired prior to inclusion to the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Gestation
Enrollment: 850 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
LGA newborns | within 24 hours after delivery
  Number (%) of large for gestational age (LGA) newborns
TRIB1 | within 24 hours after delivery
  Level of expression of TRIB1 gene
LEP | within 24 hours after delivery
  Level of expression of LEP gene
ADIPOQ | within 24 hours after delivery
  Level of expression of ADIPOQ gene
ANGPTL4 | within 24 hours after delivery
  Level of expression of ANGPTL4 gene
NR3C1 | within 24 hours after delivery
  Level of expression of NR3C1 gene

SECONDARY OUTCOMES:
Cesarian sections | within 24 hours after delivery
  Number (%) of deliveries by Cesarian sections
SGA newborns | within 24 hours after delivery
  Number (%) of small for gestationa age (SGA) newborns
Methylation of candidate genes | within 24 hours after delivery
  Levels of methylation (%) of candidate genes with confirmed differences in the expression in HUVECs isolated within 24 hours after delivery
rate of macrosomia | delivery
  birth weight ≥4000 g
birthweight | delivery
  birth weight (g)
length at birth | delivery
  length at birth (cm)
rate of stillbirth | > 20 weeks
  Foetal death in utero > 20 weeks
rate of neonatal death | 1 month after delivery
  death <1 months after delivery
rate of shoulder dystocia | delivery
  vaginal cephalic delivery in which, after the head is delivered and gentle traction proves unsuccessful, additional obstetric maneuvers are required to complete the delivery of the fetus
rate of birth trauma | delivery
  bone fracture, damage to nerves
rate of preterm birth | delivery
  babies born at <37 weeks gestational age
gestational age | delivery
  gestational age at delivery
rate of neonatal hypoglycemia | first 48 hours of age
  plasma glucose level below 2.6 mmol/L within the first 48 hours of age
rate of neonatal respiratory distress syndrome | delivery
  respiratory failure or distress
rate of jaundice | delivery
  jaundice necessitating phototherapy and/or exchange transfusion
Rate of neonates with Apgar score <7 at 5 minutes | delivery
  A measure of the health of a newborn infant done at 5 min. The newborn is given points (0, 1, 2) for heart rate, respiratory effort, muscle tone, response to stimulation and skin coloration. A score of 10 points indicates excellent health.
rate of NICU admission | within 72 hours postpartum
  neonatal intensive care unit (NICU) admission
length of stay of infants admitted to neonatal intensive care unit | up to 30 days after delivery
  length of stay of infants admitted to neonatal intensive care unit, days
cord blood C-peptide | delivery
  cord blood C-peptide levels
rate of composite neonatal outcome | delivery
  infant death, shoulder dystocia, bone fracture, and nerve palsy
rate of maternal death | within 42 days of termination of pregnancy
  death of a woman while pregnant or within 42 days of termination of pregnancy
rate of eclampsia | from 20 weeks to delivery
  generalized convulsions and/or coma
rate of placental abruption | before delivery
  premature separation of the placenta from the uterine wall before delivery
rate of postpartum hemorrhage | delivery
  requiring or offered blood transfusion or an operative procedure
rate of preeclampsia | from 20 weeks to delivery
  onset of new hypertension and proteinuria and/or end-organ dysfunction after 20 weeks of gestation
rate of gestational hypertension | from 20 weeks to delivery
  new-onset hypertension (140/90 mmHg or higher), without proteinuria after 20 weeks of gestation
rate of induction of labor | delivery
  the use of medications or other methods to bring on (induce) labour
rate of perineal trauma | delivery
  perineal or deep vaginal laceration
rate of operative vaginal delivery (vacuum extraction) | delivery
  application of vacuum to the foetal head
gestational weight gain | delivery
  Weight from preconception until last weight measured within 4 weeks before delivery.
blood pressure at admission to the birth unit | at admission to the birth unit
  blood pressure at admission to the birth unit, mm Hg
rate of maternal hypoglycemia | during pregnancy
  typical symptoms with capillary glucose <3.9 mmol/L, or, if asymptomatic, by capillary glucose <3.3 mmol/L
insulin therapy requirements | from 12 weeks to delivery
  Prescription of insulin treatment
rate of stroke | during pregnancy or within 42 days after delivery
  Maternal sudden loss of brain function due to blocked or burst blood vessels during pregnancy or postpartum.
rate of acute pulmonary oedema | During pregnancy of within 42 days after delivery
  Maternal acute pulmonary oedema
rate of cardiac arrest | During pregnancy or within 42 days after delivery
  Maternal cardiac arrest
rate of maternal respiratory arrest | During pregnancy or within 42 days after delivery
rate of maternal respiratory distress syndrome | During pregnancy or within 42 days after delivery
rate of maternal deep vein thrombosis or pulmonary embolus requiring anticoagulant therapy | During pregnancy or within 42 days after delivery
rate of maternal haemolysis | During pregnancy or within 42 days after delivery

OTHER OUTCOMES:
HbA1c | 36 week
  HbA1c level, %
fasting glucose | 36 week
  fasting plasma glucose level, mmol/L
lipid profile | 36 week
  levels of serum total cholesterol, low density lipoproteins, high density lipoproteins , triglycerides, mmol/L
glycaemic control parameters | from 12 weeks to delivery
  mean fasting and postprandial capillary glucose, adherence to target ranges via self-monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Griniva Elena, MD, PhD, Study Director — Almazov NMRC
Locations (1):
- Almazov NMRC, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hofer OJ, Martis R, Alsweiler J, Crowther CA. Different intensities of glycaemic control for women with gestational diabetes mellitus. Cochrane Database Syst Rev. 2023 Oct 10;10(10):CD011624. doi: 10.1002/14651858.CD011624.pub3. PMID 37815094